CLINICAL TRIAL: NCT01685944
Title: A Randomized, Double-blind, Placebo Controlled Study to Evaluate the Effect of Pediococcus Pentosaceus LP28 on Obesity
Brief Title: Anti-Obesity Effect of Pediococcus Pentosaceus LP28
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: eki-619
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Live Pediococcus pentosaceus LP28 (Experimental)
  Interventions: Dietary Supplement: Live Pediococcus pentosaceus LP28
- Heat-killed Pediococcus pentosaceus LP28 (Experimental)
  Interventions: Dietary Supplement: Heat-killed Pediococcus pentosaceus LP28

INTERVENTIONS:
Dietary Supplement: Live Pediococcus pentosaceus LP28
  Arms: Live Pediococcus pentosaceus LP28
Dietary Supplement: Heat-killed Pediococcus pentosaceus LP28
  Arms: Heat-killed Pediococcus pentosaceus LP28
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate efficacy of Pediococcus pentosaceus LP28 in reducing body fat and body weight in subjects with BMI 25-30 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-30 kg/m2

Exclusion Criteria:

* Taking medicines or functional food that may affect body weight or body fat
* Pregnant or nursing a child
* Participation in any clinical trial within 90 days of the commencement of the trial
* Renal or hepatic dysfunction
* Heart disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Body fat | Every 4 weeks (Overall 12 weeks)
BMI | Every day (Overall 14 weeks)
  Body weight will be measured every morning.

SECONDARY OUTCOMES:
Abdominal circumference | Every 4 weeks (Overall 12 weeks)
Serum triglyceride | Every 4 weeks (Overall 12 weeks)
Total cholesterol | Every 4 weeks (Overall 12 weeks)
LDL cholesterol | Every 4 weeks (Overall 12 weeks)
HDL cholesterol | Every 4 weeks (Overall 12 weeks)
Fasting blood glucose | Every 4 weeks (Overall 12 weeks)
Fasting insulin | Weeks 0 and 12
HOMA-R | Weeks 0 and 12
Adiponectin | Weeks 0 and 12
Leptin | Weeks 0 and 12
Resistin | Weeks 0 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Japan